CLINICAL TRIAL: NCT03050138
Title: The Prevalence of Post-Thrombotic Syndrome in Deep-Vein Thrombosis (DVT) Patients Treated With Dabigatran- a Cross-Sectional Assessment of RE-COVER Study Patients
Brief Title: Prevalence of Post-Thrombotic Syndrome in Deep-Vein Thrombosis (DVT) Patients Treated With Dabigatran
Acronym: DABI-PTS
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Ostfold Hospital Trust (Other); St. Olavs Hospital (Other); Vestre Viken Hospital Trust (Other); Sahlgrenska University Hospital (Other); Kristianstad University (Other); Jewish General Hospital (Other); McMaster University (Other)
Responsible Party: Principal Investigator, Hilde Skuterud Wik, Senior consultant in hematology, Oslo University Hospital
Other Study IDs: 2014/151
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Postthrombotic Syndrome
Keywords: Postthrombotic Syndrome; Venous Thrombosis; Quality of Life; Hemorrhage; Recurrence
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis; Hemorrhage; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dabigatran: In the RE-COVER- and RE-COVER II studies, one group of DVT and/or PE patients were randomized to receive 6 months of treatment with dabigatran (150 mg twice daily). All patients received an initial 5-7 day phase of parenteral anticoagulant treatment.
- Warfarin: In the RE-COVER- and RE-COVER II studies, the other group of DVT and/or PE patients were randomized to receive 6 months of treatment with warfarin (once daily to maintain international normalized ratio (INR) 2.0-3.0). All patients received an initial 5-7 day phase of parenteral anticoagulant treatment.

SUMMARY:
The primary objective in this cross-sectional study is to assess the prevalence of post-thrombotic syndrome (PTS) in the two treatment arms of the RE-COVER studies (warfarin versus dabigatran). PTS will be assessed by the recently developed Patient Reported Villalta (PRV) Score.

Secondary objectives: to assess in both treatment arms the

1. Prevalence of recurrent venous thromboembolism (VTE) after the discontinuation of study treatment.
2. Prevalence of PTS determined by the standard Villalta score.
3. Health related Quality of Life (HRQoL).

DETAILED DESCRIPTION:
In the RE-COVER- and RE-COVER II studies, 5109 patients with deep-vein thrombosis (DVT) and/or pulmonary embolism (PE) were randomized to receive 6 months of treatment with either dabigatran (150 mg twice daily) or warfarin (once daily to maintain international normalized ratio (INR) 2.0-3.0). All patients received an initial 5-7 day phase of parenteral anticoagulant treatment. The studies were designed as double blind, double dummy trials. RE-COVER was conducted between April 2006 to November 2008 and RE-COVER II between June 2008 and October 2010; they were completed in 2009 and 2011, respectively. A substantial number of patients are expected to have developed post-thrombotic syndrome (PTS). However, since dabigatran provides a stable level of anticoagulation throughout the treatment period and knowing that the quality of anticoagulation is an important factor in the development of PTS, we anticipate that a lower rate of PTS will be seen in the dabigatran treated patients compared to warfarin.

Patients will be interviewed and examined by the investigator if they accept to attend a clinic visit. Otherwise, a telephone interview will be performed if the patient refuses to meet up. PTS will be determined using Patient Reported Villalta (PRV) Score form. However, those who will meet for consultation will in addition be assessed for PTS by the standard Villalta score.

The primary endpoint will be the prevalence of PTS determined by Patient Reported Villalta (PRV) score. The secondary endpoints are 1- objectively verified DVT or PE after the discontinuation of treatment, 2- prevalence of PTS determined by the standard Villalta score, 3- health related quality of life (HRQOL) determined by EQ-5D (www.euroqol.org) and Venous Insufficiency Epidemiological and Economic Study quality of life and symptom (VEINES-QOL/Sym) questionnaires.

The investigators will recruit the subpopulation of patients who were included into the RE-COVER studies in the Norway, Sweden and Canada.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DVT (±PE) treated in the RE-COVER studies.
2. Signed written informed consent.

Exclusion Criteria:

1. Patients who refuse to participate
2. Deceased patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients participating in the RE-COVER- and RE-COVER II studies in Canada, Norway, Sweden, and Denmark will be invited to participate in this investigator initiated follow-up study. In the original studies patients with DVT and/or PE were randomized to receive 6 months of treatment with either dabigatran (150 mg twice daily) or warfarin (once daily to maintain international normalized ratio (INR) 2.0-3.0). All patients received an initial 5-7 day phase of parenteral anticoagulant treatment. The studies were designed as double blind, double dummy trials. RE-COVER was conducted between April 2006 to November 2008 and RE-COVER II between June 2008 and October 2010; they were completed in 2009 and 2011, respectively. The present study is a cross-sectional study.
Sampling Method: Non-Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Post-thrombotic syndrome (PTS) | April 2016 - December 2017
  The primary objective is to assess the prevalence of PTS in a subgroup of patients in the two treatment arms of the RE-COVER studies assessed by Patient Reported Villalta (PRV) Score.

SECONDARY OUTCOMES:
Recurrent venous thromboembolism | April 2016 - December 2017
  Prevalence of recurrent VTE after the discontinuation of study treatment in a subgroup of patients in the two treatment arms of the RE-COVER studies.
Post-thrombotic syndrome (PTS) determined by the standard Villalta score | April 2016 - December 2017
  Prevalence of PTS determined by the standard Villalta score in a subgroup of patients in the two treatment arms of the RE-COVER studies.
Generic health related Quality of Life (HRQoL) | April 2016 - December 2017
  Generic health related Quality of Life (HRQoL) assessed by the EQ-5D in a subgroup of patients in the two treatment arms of the RE-COVER studies.
Disease specific health related Quality of Life (HRQoL) | April 2016 - December 2017
  Disease specific health related Quality of Life (HRQoL) assessed by the VEINES-QOL/Sym score in a subgroup of patients in the two treatment arms of the RE-COVER studies.

CONTACTS AND LOCATIONS:
Overall Officials: Hilde S Wik, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (3):
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada
- Oslo University Hospital Rikshospitalet, Oslo, Norway
- Sahlgrenska Universitetssjukhuset/Östra, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Utne KK, Ghanima W, Foyn S, Kahn S, Sandset PM, Wik HS. Development and validation of a tool for patient reporting of symptoms and signs of the post-thrombotic syndrome. Thromb Haemost. 2016 Jan;115(2):361-367. doi: 10.1160/th15-04-0318. Epub 2015 Sep 17. PMID 26422814
- [Background] Schulman S, Kearon C, Kakkar AK, Mismetti P, Schellong S, Eriksson H, Baanstra D, Schnee J, Goldhaber SZ; RE-COVER Study Group. Dabigatran versus warfarin in the treatment of acute venous thromboembolism. N Engl J Med. 2009 Dec 10;361(24):2342-52. doi: 10.1056/NEJMoa0906598. PMID 19966341
- [Background] Schulman S, Kakkar AK, Goldhaber SZ, Schellong S, Eriksson H, Mismetti P, Christiansen AV, Friedman J, Le Maulf F, Peter N, Kearon C; RE-COVER II Trial Investigators. Treatment of acute venous thromboembolism with dabigatran or warfarin and pooled analysis. Circulation. 2014 Feb 18;129(7):764-72. doi: 10.1161/CIRCULATIONAHA.113.004450. Epub 2013 Dec 16. PMID 24344086